CLINICAL TRIAL: NCT03928639
Title: NHLBI Structural Heart and Valve Network Prospective Registry
Brief Title: Structural Heart and Valve Network PROSPECTIVE Registry
Status: Withdrawn | Type: Observational
Why Stopped: Due to logistical issues at Emory University enrollment never initiated.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999919087; 19-H-N087
Record Dates: First submitted 2019-04-25; First posted 2019-04-26 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Mitral Valve Regurgitation; Heart Failure; Heart Valve Disease; Tricuspid Valve Regurgitation; Aortic Valve Stenosis
Keywords: Transcatheter Aortic Valve Replacement; Mitral Valve Disease; Transcatheter Mitral Valve Replacement; Tricuspid Valve Disease; Transcatheter Mitral Valve Repair; Natural History
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure; Heart Valve Diseases; Tricuspid Valve Insufficiency; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: All patients undergoing consultation for structural and valve interventional procedures are invited to participate in this registry protocol.

SUMMARY:
Background:

Treatments for structural heart and valve disease are quickly changing. But treatment could be improved. Researchers want to gather data from people with this disease. They want to find problems and seek new ways to make treatments better.

Objective:

To find people with structural heart and valve disease with common features to study. To find flaws and patterns in procedures related to this disease. To share findings with other researchers.

Eligibility:

People ages 18 and older who are receiving care from the structural heart and valve program at the participating NHLBI structural heart disease network sites that are part of the study

Design:

Participants will be screened with their consent. This will occur when they give their standard consent for medical care.

Participants will have their data collected in the course of standard medical care. Data include:

Demographic data

Protected health data

Personally identifiable data

Medical records

Medical images. These could include X-rays, CT scans, and MRI scans.

The study could find something that would impact participants care. If this is the case, their doctors will be told.

Participants data may be shared with other researchers.

...

DETAILED DESCRIPTION:
Medical care is evolving rapidly for patients considered for treatment of structural heart and valve disease. Despite technical advances, many shortcomings remain. This research protocol allows researchers to pool medical records and imaging studies to identify problems and seek new solutions.

All patients considered for treatment at participating NHLBI structural heart and valve centers are invited to allow researchers to access their medical records repeatedly, including the results of medical procedures and imaging studies such as catheterization, CT, echocardiography, and MRI. These records, which include patient identity, will be sent to a central NHLBI database and kept confidential. Results will be used in medical publications but patient identity will be hidden.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adults age greater than or equal to 18 years.
* Receiving care from the structural heart and valve program at the participating NHLBI structural heart disease network site.
* Consent to participate in the protocol, directly, or through legally authorized representatives (LAR).

EXCLUSION CRITERIA:

- Does not consent to participate in this protocol.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing consultation for structural and valve interventional procedures, at participating NHLBI structural heart and valve centers, are invited to participate in this registry protocol.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Enrollment | Ongoing
  To identify patients with common features of interest for further analysis, for example, of specific types of complications, and identifyshortcomings and patterns in clinical structural heart and valve interventional procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Lederman, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- Emory University, Atlanta, Georgia, United States